CLINICAL TRIAL: NCT01460082
Title: Endothelial Dysfunction and Systemic Inflammation in Patients With Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Endothelial Dysfunction in Acute Exacerbations of Chronic Obstructive Pulmonary Disease (COPD)
Acronym: EDAECOPD
Status: Completed | Type: Observational
Sponsor: LudwLudwig Boltzmann Institute for COPD and Respiratory Epidemiology (Network)
Responsible Party: Principal Investigator, Matthias Urban, M.D., Study coordinator, LudwLudwig Boltzmann Institute for COPD and Respiratory Epidemiology
Other Study IDs: EDAECOPD
Record Dates: First submitted 2011-10-25; First posted 2011-10-26 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Inflammatory Disease; Endothelial Dysfunction
Keywords: chronic obstructive pulmonary disease; acute exacerbation; endothelial dysfunction; flow mediated dilation; systemic inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exacerbation: The study sample will consist of patients admitted to the hospital because of an acute exacerbation of COPD

SUMMARY:
The purpose of the study is to determine a possible association between the clinical entity of exacerbation, markers of systemic inflammation and endothelial dysfunction in patients with COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a chronic inflammatory disease of the lungs; however, there is cumulating data suggesting that the inflammatory reaction associated with COPD is not restricted to the lungs but has systemic effects. Patients with COPD have increased cardiovascular morbidity and mortality. The suspected link between increased cardiovascular mortality and systemic inflammation is endothelial dysfunction, which in turn is caused by impaired activity of NO. Endothelial dysfunction has been demonstrated in patients with COPD. Furthermore there is a close correlation between endothelial dysfunction in coronary and peripheral vessels, which allows assessing flow-mediated dilation (FMD) in the brachial artery via high resolution ultrasound as an early predictor of atherosclerosis. Moreover, systemic inflammatory markers correlate with endothelial dysfunction in patients with stable COPD.

Exacerbations of COPD are episodes of worsening symptoms characterized by increased airway and systemic inflammation. If systemic inflammation is a cause of endothelial dysfunction in COPD, endothelial function would be suspected to be further impaired during exacerbation and recover thereafter. The purpose of this study is to determine a possible association between the clinical entity of exacerbation, markers of systemic inflammation and endothelial dysfunction in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* presence of COPD according to standard criteria
* acute exacerbation of COPD according to recommended international criteria
* over 40 years of age
* history of at least 10 py

Exclusion Criteria:

* pneumonia
* history or signs of congestive heart failure,
* acute myocardial infarction
* thoracotomy incl. resection of lungtissue
* interstitial lung disease
* acute or chronic renal failure
* active malignancy
* autoimmune disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD diagnosed according to standard criteria in the state of acute exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
change of endothelial dysfunction (impaired vasomotor reactivity due to shaer stress) confirmed by non-invasive measurement of flow mediated dilation (FMD) 6-8 weeks after acute exacerbation of COPD | Baseline, Week 6-8

SECONDARY OUTCOMES:
change of systemic inflammation 6-8 weeks after COPD-exacerbation confirmed by inflammatory markers such as interleukin-6 (IL-6), fibrinogen levels, and C-reactive protein (CRP) levels | baseline, week 6-8

CONTACTS AND LOCATIONS:
Overall Officials: Georg C Funk, M.D., Principal Investigator — 1. Department of Respiratory and Critical Care Medicine and Ludwig Boltzmann Institute for COPD, Otto-Wagner Hospital, Vienna, Austria
Locations (1):
- 1.Department of Respiratory and Critical Care Medicine and Ludwig Boltzmann Institute for COPD, Otto-Wagner Hospital, Vienna, Vienna, Austria